CLINICAL TRIAL: NCT07295067
Title: An Exploratory Study on the Use of Intrathecal Injection of Human Autologous Mesenchymal Stromal Cells Derived Extracellular Vesicles for the Treatment of Syringomyelia
Brief Title: Extracellular Vesicles for the Treatment of Syringomyelia
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Xuanwu Hospital, Beijing (Other)
Collaborators: Yisaier Medical Technology (shan xi) Co., Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XWhUC-MSCs-EV
Record Dates: First submitted 2025-11-19; First posted 2025-12-19 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-12

CONDITIONS: Syringomyelia
Keywords: syringomyelia; spinal cord injury; mesenchymal stromal cell; extracellular vesicle
MeSH Terms: conditions — Syringomyelia; Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exosomes group (Experimental): Patients in this arm will receive exosomes derived from human umbilical cord blood mesenchymal stem cells as a Intrathecal injection, administered once a month, for a total of three months.
  Interventions: Drug: Exosomes group

INTERVENTIONS:
Drug: Exosomes group — Exosomes derived from human umbilical cord blood mesenchymal stem cells for Intrathecal injection (administered once a month, for a total of three months, based on the recommended dose during the dose-escalation phase).

SUMMARY:
This is a open-label, single-arm, dose escalation phase I clinical trial. The goal of this clinical trial is to evaluate the safety and preliminary efficacy of Intrathecal injection human umbilical cord-derived mesenchymal stromal cell-derived extracellular vesicle (hUC-MSC-sEV) in syringomyelia.

DETAILED DESCRIPTION:
This is a open-label, single-arm, dose escalation phase I clinical trial. The study will consist of one part: Part 1 will be a dose-escalation study.

A traditional 3+3 dose-escalation design will be implemented in Part 1. Cohort 1 will receive low-dose1×1011particles; Cohort 2 will receive middle-dose2×1011particles; and Cohort 3 will receive high-dose3×1011particles. (Cohort 1 to Cohort 3 will receive a dose of 2 ml per lumbar puncture, administered once a month, for a total of three months.) If no dose-limiting toxicities (DLTs) are observed for 2 weeks after the administration of the first Intrathecal injection, a new cohort will be enrolled at the next planned dose level. If DLTs are observed in one participant in the cohort, an additional three participants will be treated at the same dose level. Dose escalation will be stopped if DLTs are observed in more than 33% of the participants.

ELIGIBILITY:
Inclusion Criteria:

* Patients whose MR revealed that syrinx have shrunk after surgery for a year but whose clinical spinal cord symptoms have not improved.
* Patients whose MR revealed that syrinx spontaneously resolution under conservative observation, but whose clinical spinal cord symptoms have not improved.
* Age: 18-70 years, inclusion of both genders;

Exclusion Criteria:

* 1. Those with diabetes, heart disease, or impaired liver or kidney function; 2. Those with other diseases such as brainstem tumors and spinal cord tumors; 3. Infected individuals with lumbar puncture sites; 4. Those with previous or detected abnormalities in the heart; 5. Those who have autoimmune diseases and need to be treated with immunosuppressants; 6. Those who are allergic to the research drugs; 7. Have participated in other interventional clinical studies or received other cell therapies (excluding blood transfusion) within the past three months; 8. Those who are unconscious, unable to express subjective discomfort symptoms and unable to cooperate with neurological function tests, those who have been receiving drug treatment for a long time and do not cooperate with the treatment plan; 9. Pregnant women, women who are breastfeeding and those planning to become pregnant; 10. Serological tests (HBsAg, anti-HCV, anti-HIV, TP-Ab) are positive; 11. Other circumstances where the researcher deems the patient unsuitable to participate in this study (including but not limited to not meeting the treatment that benefits the patient the most, poor patient compliance, abnormal laboratory test indicators that cannot be accepted, etc.).

Rejection Criteria:

misdiagnosis; use of any medication that may significantly impact the assessment accuracy of hUC-MSC-sEV engraftment; absence of any evaluation outcome at any time point during the follow-up period

Cessation Criteria:

individual wishes of the subjects; occurrence of any hUC-MSC-sEV-associated serious adverse event (SAE) that may aggravate neurological dysfunction, or require prolongation of existing hospitalization, or need hospital readmission, or impair consciousness, or be life-threatening, or even lead to death in any subject; detection of any major mistake in the present protocol during the implementation of this clinical trial; the national administration agency requires the clinical trial to be halted

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2025-12-23 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants who experienced dose-limiting Toxicities (DLTs) | 24 hours, 4±1 Weeks, 8±1 Weeks,12±1 Weeks
  DLTs related to hUC-MSC-sEV include adverse events of grade 3 or higher (including significant clinical laboratory findings) that are possibly, likely, or definitely related to the study drug, accompanied by clinical symptoms and requiring medical treatment within 14 days of administration. Adverse events are graded according to the Common Terminology Criteria for Adverse Events Version 5.0 (CTCAE 5.0).

SECONDARY OUTCOMES:
American Spinal Injury Association(ASIA) Score | 4±1 Weeks, 8±1 Weeks,12±1 Weeks, 12±1 months
  American Spinal Injury Association(ASIA) Score for evaluating the spinal cord function， degree of the spinal cord function, motor1-100, sensory 1-224, higher scores mean a better outcome
Klekamp and Sammi syringomyelia scale | 4±1 Weeks, 8±1 Weeks,12±1 Weeks, 12±1 months
  for evaluating the spinal cord function, each score 1-5, higher scores mean a better outcome
Incidence of severe adverse events | 4±1 Weeks, 8±1 Weeks,12±1 Weeks
  The proportion of patients who experienced severe adverse events.
Time to event (death, tracheostomy, and permanent assisted mechanical ventilation) | up to 12 months
  The number of time-to-event outcomes.
modified Japanese Orthopaedic Association Scores (mJOA) | 4±1 Weeks, 8±1 Weeks,12±1 Weeks, 12±1 months
  Motor function， sensory， bladder function；for evaluating the spinal cord function；0-17， higher scores mean a better outcome
xuanwu syringomyelia scale | 4±1 Weeks, 8±1 Weeks,12±1 Weeks, 12±1 months
  for evaluating the spinal cord function, for evaluating the spinal cord function；0-18， higher scores mean a worse outcome
improvement or resolution of the syrinx | 4±1 Weeks, 8±1 Weeks,12±1 Weeks, 12±1 months
  improvement in size.

OTHER OUTCOMES:
Change from baseline in the blood and csf markers. | 4±1 Weeks, 8±1 Weeks,12±1 Weeks
  A number of blood and csf markers will be examined.
Change from baseline in the neuroimaging indices. | 4±1 Weeks, 8±1 Weeks,12±1 Weeks
  Neuroimaging indices include DTI, DTI-ALPS.
Change from baseline in the Electrophysiological indices. | 4±1 Weeks, 8±1 Weeks,12±1 Weeks
  Electrophysiological indices include EMG.
Change from baseline in the neuroimaging indices. | 4±1 Weeks, 8±1 Weeks,12±1 Weeks
  Neuroimaging indices include QSM.
Change from baseline in the Electrophysiological indices. | 4±1 Weeks, 8±1 Weeks,12±1 Weeks
  Electrophysiological indices include Somatosensory evoked potential .
Change from baseline in the Electrophysiological indices. | 4±1 Weeks, 8±1 Weeks,12±1 Weeks
  Electrophysiological indices include Motor Evoked Potential.

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital, Beijing, Beijing City, China

IPD SHARING:
Plan to Share IPD: No
The study will not share individual participant data to other researchers.

REFERENCES:
- [Background] Yuan C, Du Y, Yao Q, Zhang C, Zhang L, Liu Z, Wang K, Duan W, Wang Z, Wang X, Zeng G, Wu H, Chen Z, Heiss JD, Guan J, Jian FZ. Natural history of Chiari I malformation-syringomyelia: longitudinal cohort study. J Neurol Neurosurg Psychiatry. 2025 Nov 13;96(12):1204-1214. doi: 10.1136/jnnp-2025-336023. PMID 40675800
- [Background] Krause M, Gburek-Augustat J, Grafe D, Metzger R, Ginzel M, Griessenauer CJ, Grassner L, Weghuber D, Gradl J, Auer D, Schally T, Rund S, Kals C, Folie C, Bayer E, Gimona M, Rohde E. First-In-Human Application of Human Umbilical Cord-Derived Extracellular Vesicles in Tethered Spinal Cord Release Surgery. J Extracell Vesicles. 2025 Jun;14(6):e70104. doi: 10.1002/jev2.70104. PMID 40536443
- [Background] Vaquero J, Zurita M, Rico MA, Aguayo C, Fernandez C, Rodriguez-Boto G, Marin E, Tapiador N, Sevilla M, Carballido J, Vazquez D, Garcia-Olmo D, Guadalajara H, Leon M, Valverde I; Neurological Cell Therapy Group From Puerta De Hierro-Majadahonda Hospital. Cell therapy with autologous mesenchymal stromal cells in post-traumatic syringomyelia. Cytotherapy. 2018 Jun;20(6):796-805. doi: 10.1016/j.jcyt.2018.04.006. Epub 2018 May 18. PMID 29784434
- [Background] Li M, Wang X, Qi B, Cui S, Zheng T, Guan Y, Ma L, Liu S, Li Q, Chen Z, Jian F. Treatment of Syringomyelia Characterized by Focal Dilatation of the Central Canal Using Mesenchymal Stem Cells and Neural Stem Cells. Tissue Eng Regen Med. 2024 Jun;21(4):625-639. doi: 10.1007/s13770-024-00637-1. Epub 2024 Apr 5. PMID 38578425